CLINICAL TRIAL: NCT06114797
Title: Chamomile Effect on Xerostomia Associated With End-stage Renal Disease in Elderly: A Randomized Clinical Trial With a Biochemical Assessment
Brief Title: Chamomile Effect on Xerostomia Associated With End-stage Renal Disease in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Asmaa Aboubakr, Lecturer Assistant, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDASU-Rec IR 042308
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Xerostomia Due to Hyposecretion of Salivary Gland
Keywords: chamomile; Nitric oxide; hemodialysis; xerostomia; salivary flow rate
MeSH Terms: conditions — Xerostomia | interventions — Chamomile extract

STUDY DESIGN:
Intervention Model Description: Treatment protocol (for the intervention group):
  * Chamomile will topically be applied to the oral mucosa as oral rinse based on the Morales-Bozo I et al., (2017) administration protocol.
  * Based on this protocol, patients will have oral rinses 3 times per day.
  * Patients will be instructed to perform chamomile rinses in the oral mucosa.
  * Patients will be instructed not to swallow the chamomile oral rinse.
  The control group (placebo):
  Patients in the control arm followed the same protocol with normal saline rinses. As stated by Kim JO and Kim NC, 2014, that use of 4% hypertonic saline solution mouthwash by elderly provided better oral health by decreasing xerostomia, oral tongue plaque, halitosis, and the number of oral bacteria.
  So the patients in the control group will be benefited from the saline oral rinse.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants in both groups will not recognize the type of applied treatment whether it is saline mouthwash or chamomile mouthwash.
  Outcome assessor will not know whether the patients they are assessing are from the control or the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chamomile mouthwash interventional arm in elderly patients having end-stage renal disease. (Active Comparator): * Chamomile was topically applied to the oral mucosa as oral rinse.
  * Based on this protocol, patients were had oral rinses 3 times per day.
  * Patients were instructed to perform chamomile rinses in the oral mucosa.
  * Patients were instructed not to swallow the chamomile oral rinse.
  Interventions: Other: Chamomile
- Saline mouthwash control group in elderly patients having end-stage renal disease. (Placebo Comparator): Patients in the control arm followed the same protocol with normal saline rinses. As stated before, that use of 4% hypertonic saline solution mouthwash by elderly provided better oral health by decreasing xerostomia, oral tongue plaque, halitosis, and the number of oral bacteria.
  So the patients in the control group were benefited from the saline oral rinse.
  Interventions: Other: Saline mouthwash

INTERVENTIONS:
Other: Chamomile — * Chamomile was topically applied to the oral mucosa as oral rinse.
  * Based on this protocol, patients had oral rinses 3 times per day.
  * Patients were instructed to perform chamomile rinses in the oral mucosa.
  * Patients were instructed not to swallow the chamomile oral rinse.
  Arms: Chamomile mouthwash interventional arm in elderly patients having end-stage renal disease.
Other: Saline mouthwash — Saline mouthwash was used by elderly patients in the control arm.
  Arms: Saline mouthwash control group in elderly patients having end-stage renal disease.

SUMMARY:
Background and Objectives: Chronic hemodialysis causes changes in blood chemistry as well as dry mouth, due to removal of excess fluids. Dry mouth is due to hyposalivation or change in saliva composition. Many herbal medicines have been used as treatment options. Since the chamomile was suggested as a potent oral moisturizer by previous studies that have been done in this field. Therefore, the investigators decided to assess the effect of chamomile oral rinse on the SXI score, salivary nitric oxide level, salivary flow rate, OHIP-14, serum creatinine and blood urea levels in elderly patients on chronic hemodialysis.

Material and Methods: It is an interventional randomized controlled clinical trial with a biochemical assessment. A chamomile, and placebo mouthwashes were provided to eighty-eight elderly participants with end-stage renal disease suffering from xerostomia. Patients were divided into 2 equal groups who used either the chamomile or placebo mouthwash for one month. The SXI score and salivary flow rate were evaluated for both groups at different intervals (baseline, 1 week, and 1 month). While salivary NO levels, OHIP-14, serum creatinine and blood urea levels evaluated at baseline and after one month only.

DETAILED DESCRIPTION:
A double-blind (interventional) cross-sectional clinical trial was performed on 88 participants in the hemodialysis center at Benha university. The inclusion criteria were both genders above 30 years of age with ESRD and complaints of dry mouth sensation. The exclusion criteria were significant salivary gland damage (for example, due to anticancer medication), radiotherapy or chemotherapy history, and allergies).

Bottles containing chamomile mouthwash or the placebo (A or B) were tagged by a reliable person outside the research group and placed inside an opaque envelope along with the questionnaires. Each patient received two envelopes containing a bottle (A & B) and a questionnaire. The results were analyzed exclusively by a statistics consultant at the end of the research. The patients were asked to express their sensation of dry mouth using subjective dry mouth score.

The Summated Xerostomia Inventory (SXI) (Thomson et al., 2011; Frigaard et al., 2023):

ESRD patients who met the eligibility criteria were asked about their subjective severity of xerostomia using SXI score where the patient evaluates the frequency of complaints regarding five statements all recorded at 3 different intervals (at baseline- after 2 weeks- after 1 month).

Salivary flow rate: Eating and talking were prohibited during the time of collection. Unstimulated whole saliva was collected for 5 min by spitting method. The collection was timed, so that flow rate (mL/min) could be measured.

The Oral Health Impact Profile (OHIP-14) utilizes a scale with five categories (1 = never, 2 = hardly ever, 3 = occasionally, 4 = fairly often, and 5 = very often) that was evaluated after one month in both groups. A lower score in any of the five categories indicates higher satisfaction (Al-Zubeidi et al., 2012).

Serum creatinine and blood urea levels were assessed at baseline and after one month in both groups.

Nitric oxide levels were determined by Nitric Oxide Assay Kit (Colorimetric) using Griess reaction: The Bio Diagnostic Nitrite Assay Kit provides an accurate and convenient method for measurement of endogenous nitrite concentration as an indicator of nitric oxide production in biological fluids. It depends on the addition of Griess Reagents which convert nitrite into a deep purple azo compound, photometric measurement of the absorbance due to this azo chromophore accurately determines NO2 - concentration.

ELIGIBILITY:
Inclusion Criteria:

* Both genders, aged above 65 years.

  * All patients must be clinically diagnosed of ESRD undergoing hemodialysis.
  * Patients on hemodialysis ≥ 3 months (Bots et al., 2005).
  * All patients must have complaint of xerostomia.
  * Patients must be able to make reliable decision or communications.

Exclusion Criteria:

* - Smoking, Alcohol.
* Patient with history of any serious illness as malignancy, who undergo kidney transplant.
* Patients with any autoimmune disease.
* Vulnerable groups such as prisoners, mentally and physically handicapped individuals.

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Both genders with end-stage renal disease
Enrollment: 88 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
The Summated Xerostomia Inventory (SXI) | one month
  subjective severity of xerostomia using SXI score where the patient evaluates the frequency of complaints regarding five statements. Each statement has three possible replies: never, occasionally, or often, with scoring 1, 2, and 3, respectively. The SXI has a score range from (5 to 15), where a maximum score indicates severe problems related to dry mouth

SECONDARY OUTCOMES:
Increase in unstimulated Salivary Flow Rate (ml/min) | one month
  Unstimulated whole saliva was collected for 5 min by spitting method. The collection was timed, so that flow rate (mL/min) could be measured. The normal unstimulated salivary flow rate is approximately 0.3-0.4 mL/min. A diagnosis of hyposalivation is made when the unstimulated salivary flow rate is ≤0.1 mL/min.
  Time Frame: baseline, 2 weeks and 4 weeks after intervention ] The outcome measure will be measured before and 2 and 4 weeks after continuous usage of chamomile mouth rinse (for at least 5 days per week)
Increase in salivary Nitric oxide levels (mmol/L) using clorimetric determination method | one month
  Increase in salivary Nitric oxide levels (mmol/L) using clorimetric determination method [ Time Frame: baseline and 4 weeks after intervention] The outcome measure will be measured before and 4 weeks after continuous usage of chamomile mouth rinse (for at least 5 days per week).
The Oral Health Impact Profile (OHIP-14) questionnaire | one month
  (OHIP-14) utilizes a scale with five categories (1 = never, 2 = hardly ever, 3 = occasionally, 4 = fairly often, and 5 = very often) that was evaluated after one month in both groups. A lower score in any of the five categories indicates higher satisfaction
Serum creatinine and blood urea levels | one month
  Kidney clinical parameters to evaluate the renal function, higher values are the worst, and lower values are the best.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
will not share my raw data

REFERENCES:
- [Background] Afsaneh Abadi P, Koopaie M, Montazeri R. Comparison of salivary nitric oxide and oral health in diabetic patients with and without xerostomia. Diabetes Metab Syndr. 2020 Jan-Feb;14(1):11-15. doi: 10.1016/j.dsx.2019.11.014. Epub 2019 Nov 25. PMID 31809967
- [Background] Alam F, Islam MA, Gan SH, Khalil MI. Honey: a potential therapeutic agent for managing diabetic wounds. Evid Based Complement Alternat Med. 2014;2014:169130. doi: 10.1155/2014/169130. Epub 2014 Oct 15. PMID 25386217
- [Background] Anil S, Vellappally S, Hashem M, Preethanath RS, Patil S, Samaranayake LP. Xerostomia in geriatric patients: a burgeoning global concern. J Investig Clin Dent. 2016 Feb;7(1):5-12. doi: 10.1111/jicd.12120. Epub 2014 Sep 1. PMID 25175324
- [Background] Bardow A, Nyvad B, Nauntofte B. Relationships between medication intake, complaints of dry mouth, salivary flow rate and composition, and the rate of tooth demineralization in situ. Arch Oral Biol. 2001 May;46(5):413-23. doi: 10.1016/s0003-9969(01)00003-6. PMID 11286806
- [Background] Belcher J. Dressings and healing with honey. Br J Nurs. 2014 Mar 27-Apr 9;23(6):S22. doi: 10.12968/bjon.2014.23.Sup6.S22. PMID 24690746
- [Background] Bots CP, Brand HS, Veerman EC, Korevaar JC, Valentijn-Benz M, Bezemer PD, Valentijn RM, Vos PF, Bijlsma JA, ter Wee PM, Van Amerongen BM, Nieuw Amerongen AV. Chewing gum and a saliva substitute alleviate thirst and xerostomia in patients on haemodialysis. Nephrol Dial Transplant. 2005 Mar;20(3):578-84. doi: 10.1093/ndt/gfh675. Epub 2005 Jan 21. PMID 15665029